CLINICAL TRIAL: NCT06862908
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of IBI362 in Subjects With HFpEF（Heart Failure With Preserved ejectIon Fraction）or HFmrEF（Heart Failure With Mildly Reduced Ejection Fraction）Combined With Obesity
Brief Title: A Study of IBI362 in Subjects With HFpEF or HFmrEF Combined With Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362G201
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Heart Failure With Preserved Ejection Fraction (HFPEF); Heart Failure With Mildly Reduced Ejection Fraction
MeSH Terms: conditions — Obesity | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 4.0mg (Experimental)
  Interventions: Drug: IBI362
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- IBI362 6.0mg (Experimental)
  Interventions: Drug: IBI362

INTERVENTIONS:
Other: placebo — placebo administered subcutaneously(SC), once a week
  Arms: placebo
Drug: IBI362 — IBI362 administered subcutaneously(SC), once a week
  Arms: IBI362 4.0mg; IBI362 6.0mg

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled clinical study to evaluate the efficacy and safety of IBI362 in Chinese subjects with heart failure with ejection fraction retention/mild ejection fraction reduction (HFpEF/HFmrEF) combined with obesity (BMI≥28kg/㎡). This study will enroll about 141 NYHA Class II-III HFpEF/HFmrEF subjects combined with obesity. Eligible participants will be randomly assigned to IBI362 4 mg, IBI362 6 mg, or placebo at a ratio of 1:1:1, randomized by concomitant atrial fibrillation during screening (history/screening ECG).

The trial period includes a 2-week screening period, a 52-week double-blind treatment period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 at the time of signing the informed consent.
2. BMI≥28kg/m2.
3. NYHA class II-III.
4. There were no hospitalizations due to heart failure at screening visit (V1) to randomized visit (V2).
5. KCCQ-CSS score < 80 during the screening period and before randomization.
6. Medication for chronic diseases: If used before screening, the dose should be stable for ≥4 weeks; If not used before screening, the drug should also be stopped for ≥4 weeks.
7. The women of childbearing potential（WOCBP） agrees to use the contraceptive method prescribed in this protocol for the entire study period and for 3 months after the final treatment. Pregnancy test results for fertile women during the screening period must be negative. Female subjects should not breastfeed.
8. Voluntarily sign the informed consent form, and be willing to strictly abide by the requirements and restrictions of the informed consent form and the protocol throughout the study period, including but not limited to: maintaining a stable diet and exercise lifestyle, injecting the study drugs as planned, and keeping a study diary.

Exclusion criteria:

1. myocardial infarction, stroke, or transient ischemic attacks, hospitalization for acute heart failure requiring any ventilatory and circulatory support devices (such as IABP ,I MPELLA, ECMO, CRRT, etc.) within 3 months before screening.
2. Unstable angina pectoris or HF decompensation requiring IV diuretics, IV inotropes, or IV vasodilators within 30 days before screening.
3. Poorly controlled hypertension at the screening stage, with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg. Or systolic blood pressure < 90mmHg during screening.
4. Had previously undergone or planned to undergo bariatric surgery during the study period.
5. The presence of endocrine diseases or medical history that may significantly affect body weight.
6. Previous diagnosis of type 1 diabetes or specific type diabetes.
7. Use of GLP-1R agonists or glucagon receptor (GLP-1R/GCGR) agonists or GIPR (Glucagon dependent insulinotropic polypeptide) within 3 months before screening receptor) /GLP-1R agonist or GIPR/GLP-1R/GCGR agonist; Participants who stopped using these drugs more than 3 months prior to screening due to lack of efficacy or intolerance should also be excluded.
8. Use of insulin in the 3 months prior to screening to control diabetes, except for short-term (cumulative ≤14 days) use of insulin in acute conditions, such as acute illness, hospitalization, or elective surgery. The last insulin treatment was less than 14 days from the screening date.
9. History of medullary thyroid carcinoma, multiple endocrine neoplasia (MEN) 2A or 2B or family history.
10. Clinically significant gastric empting abnormalities (such as severe diabetic gastroparesis, gastric pyloric obstruction, etc.) or gastrointestinal surgery.
11. Active or untreated malignancies were present within 5 years prior to screening, or clinical malignancies were in remission (except in subjects with no recurrence after surgery for basal cell and squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the prostate, or papillary thyroid carcinoma).
12. A history of atopic reactions (clinical manifestations of severe or multiple allergies) or a history of clinically significant multiple or severe drug allergies, or intolerance to local glucocorticoids, Or severe post-treatment hypersensitivity reactions (including but not limited to erythema multiforme, linear immunoglobulin A dermatitis, toxic epidermal necrolysis, anaphylaxis, angioedema, or exfoliative dermatitis).
13. History of organ transplantation (except corneal transplantation, autologous skin transplantation), or preparing to receive organ transplantation.
14. The investigators identified major surgeries that might be planned during the study period that would affect the participants' ability to walk.
15. Past suicidal thoughts or behaviors.
16. The investigator believes that the subjects are not suitable to participate in the study because of any other factors (including previous serious mental illness) that may affect the efficacy, safety evaluation or compliance of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-24 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) | From baseline (week 0) to week 36
  The KCCQ is a standardized 23-item, self-administered instrument that quantifies heart failure symptoms (frequency, severity, and recent change), physical limitation, quality of life, and social limitation. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Body weight change from baseline at week 36 | From baseline (week 0) to week 36

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) | From baseline (week 0) to end of treatment (week 52)
  The KCCQ is a standardized 23-item, self-administered instrument that quantifies heart failure symptoms (frequency, severity, and recent change), physical limitation, quality of life, and social limitation. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. KCCQ-CSS includes the symptom and physical limitation domains of the KCCQ. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Body weight change from baseline at week 52 | From baseline (week 0) to end of treatment (week 52)
Incidence, severity, and association with study drugs of adverse events | From baseline (week 0) to end of treatment (week 52)
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 52)
Change in Diastolic Blood Pressure(DBP) | From baseline (week 0) to end of treatment (week 52)
Change in ECG heart rate | From baseline (week 0) to end of treatment (week 52)
  The electrocardiogram is performed by a 12-lead electrocardiogram machine
Change in N terminal pro B type natriuretic peptide（NT-proBNP） | From baseline (week 0) to end of treatment (week 52)
Change in hypersensitive C-reactive protein（hsCRP） | From baseline (week 0) to end of treatment (week 52)
Occurrence of serum anti-iBI362 antibody (ADA) before and after administration | From baseliFrom baseline (week 0) to end of treatment (week 52)ne (week 0) to week 52
Occurrence of neutralizing antibody (NAb) before and after administration | From baseline (week 0) to end of treatment (week 52)
Pharmacokinetics (PK): Maximum Concentration (Cmax) of IBI362 | From baseline (week 0) to end of treatment (week 52)
PK: Area Under the Concentration Versus Time Curve (AUC) of IBI362 | From baseline (week 0) to end of treatment (week 52)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China